CLINICAL TRIAL: NCT06480916
Title: Study of the Value of Maternal-fetal Transfers and Their Complexity of Their Implementation
Acronym: TRANSFERT
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-04Obs-CHRMT
Record Dates: First submitted 2024-06-19; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Maternal-Fetal Relations
Keywords: maternal-fetal transfer; care organization; patient pathway; maternity hospital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Maternal-fetal transfers — Prospective and consecutive inclusion of all maternal-fetal transfers during the study period. The teams at the sending and receiving maternity units will complete study-related questionnaires to describe the conditions of the transfer and the outcome of the pregnancy. The study in no way alters the way parturients are cared for.

SUMMARY:
It is an observational, descriptive, prospective, multicenter study of 8 maternity units in Lorraine and Champagne-Ardenne, aimed at comparing the percentage of "avoidable" maternal-fetal transfers (MFTs), defined as transfers in which the delivery finally meets the acceptance criteria of the sending maternity unit, according to the obstetrical indications for these MFTs.

DETAILED DESCRIPTION:
Over the past year, an audit carried out on the Mercy maternity unit, covering 130 transfers to the Nancy regional maternity hospital, showed that patients transferred for threat of premature delivery (MAP) with a cervix > 15 mm do not give birth at the receiving maternity unit, but return home after 48 hours' hospitalization.

When maternal-fetal transfer (MFT) is requested, numerous calls are made to private ambulance services, and in the end, many emergency rapid response units (SMUR) are called out, requiring a major human, logistical and time investment for a questionable benefit to the patient. Tensions in terms of logistics (lack of ambulance, SMUR) and human resources (lack of personnel) can, conversely, compromise good care of the parturient.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman cared for in a participating maternity unit
* Over 18 years of age
* Requested for maternal-fetal transfer (finally performed, or not)

Exclusion Criteria:

* missing data on transfer outcome

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Maternal-fetal transfers (MFTs) for threatened premature delivery
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
The percentage of "avoidable" maternal-foetal transfer (MFT) | after delivery, up to 6 weeks after the maternal-foetal transfer
  The main evaluation criterion is "avoidable" maternal-foetal transfer (MFT), i.e. resulting in a delivery that met the acceptance criteria of the original maternity hospital

SECONDARY OUTCOMES:
Obstetrical indication for maternal-foetal transfer (MFT) | Up to 48 hours after the maternal-foetal transfer
  as documented in the patient file
Organizational arrangements for maternal-foetal transfer | Up to 6 months after inclusion of a maternity unit in the study
  Organizational arrangements for maternal-foetal transfer in the various centers, assessed by a specific questionnaire sent to maternity units.

CONTACTS AND LOCATIONS:
Overall Officials: Laetitia HONORE-ROUGE, MD, Principal Investigator — CHR Metz Thionville Hopital Femme Mère Enfant
Locations (8):
- France (8):
  - Hopital Maillot, Briey
  - Maternité CH Léon Bourgeois, Châlons-en-Champagne
  - CHR Metz Thionville Hopital Femme Mère Enfant, Metz
  - Maternité - Hôpital Maurice Camuset, Romilly-sur-Seine
  - Clinique Saint Nabor, Saint-Avold
  - Matérnité Saint Dizier, Saint-Dizier
  - CHR Metz-Thionville Hopital Bel Air, Thionville
  - Hopital Saint Nicolas, Verdun

IPD SHARING:
Plan to Share IPD: No